CLINICAL TRIAL: NCT02654574
Title: Comparison of Two Modes of Administration of the IADL Questionnaire
Brief Title: Comparison of Two Modes of Administration of the IADL Questionnaire, Assessing the Level of Functional Autonomy of Patients to Carry Out the Tasks of Daily Living: Randomized Controlled Trial Among Patients of a Memory Clinic
Acronym: IADL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014-867; 2014-A00446-41 (Other: ANSM)
Record Dates: First submitted 2016-01-11; First posted 2016-01-13 (Estimated); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer's Disease; Dementia Disorders
Keywords: Alzheimer's disease or related disorders; Functional autonomy level; Lawton Instrumental Activities of Daily Living; The Functional autonomy level
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Face-to-face collection followed by collection by phone (Experimental): Reference procedure i.e IADL collected during a face-to-face interview at the Memory Clinic, followed by the collection of IADL by phone, one month later.
  Interventions: Other: IADL administration by phone
- Collection by phone followed by face-to-face collection (Experimental): Collection of IADL by phone, followed by the collection of the IADL questionnaire using the reference procedure i.e IADL collected during a face-to-face interview at the Memory Clinic, one month later.
  Interventions: Other: IADL administration by phone

INTERVENTIONS:
Other: IADL administration by phone — The administration of IADL questionnaire by phone consists of a collection of answers given by the caregiver during the interview with the research nurse, trained for this procedure. This method of procurement will be standardized with a listing support for the phone interview to obtain the same conditions for collection of data from a caregiver to another. Questions will be asked in the same order than the questionnaire collected with the reference procedure i.e. face-to-face interview at the Memory Clinic. The IADL questionnaires in paper format used during the ace-to-face interview and by phone will be identical.

SUMMARY:
In France, about 1 million people 65 and older are diagnosed with dementia syndrome characterized by cognitive decline and impairment of functional capacity. The assessment of the level of functional autonomy is therefore an essential step in monitoring patients in Memory Clinic and can be estimated by the Lawton IADL questionnaire, assessing the patients' ability to perform daily tasks.

In the Memory Clinic, the first estimate of the level of patient autonomy is achieved during a face-to-face interview between their primary caregiver and a nurse, using the IADL questionnaire. This assessment should be renewed every year. The IADL questionnaire is part of the information that the memories consultations shall transmit to the Alzheimer's National Bank (BNA).

However, current practice has shown that the systematic collection is problematic in the organization of Memory Clinic. It is thus expected to collect this questionnaire by phone in order to measure changes in the level of autonomy during the disease, and improve the completeness of this collection. A study is conducted with the main objective to measure the reliability of the assessment of IADL questionnaires conducted during a telephone interview with the caregiver of the patient, in comparison to the reference mode: the face-to-face interview with the caregiver.

Materials and methods The experimental design of the study will be a randomized crossover trial (crossover), including 394 patients divided into two branches. In the first part, the collection of the IADL questionnaire will be performed according to the reference method in the consultation (face-to-face interview with the nurse), the measurement will be repeated at 1 month intervals by phone. In the second part the sequence of execution modes will be reversed. The reliability of the measurement of the level of autonomy will be studied by comparing repeated measurements based on handover modes. The correspondence between the repeated measures will also be considered in terms of patient characteristics. The feasibility of administration of the questionnaire by phone mode will be evaluated.

Expected results The mode of administration by phone should allow to obtain a reliable measurement of the level of patient autonomy when the administration is carried out in a standardized way. The study should also identify patients and situations for which this method of administration by phone may be appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Patients received for the first time at the Memory Clinic,
* Patients living at home
* Patients accompanied by a caregiver,
* Patients and caregivers agreeing to participate in the study.

Exclusion Criteria:

* Patients whose caregivers did not wish to participate in the study,
* Patients living in institutions or nursing homes,
* Patients whose caregivers did not have or did not provide a telephone contact,
* Patients for who the health status would require institutionalization during the period of the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2014-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Degree of agreement (concordance) of the overall level of functional autonomy measured with two ways (face-to-face interview and by phone) | 1 month
  The degree of agreement (concordance) of the overall level of autonomy will be measured between the two modes administration of the IADL questionnaire.
  The level of independence (or dependence) will be evaluated from the scale of instrumental activities of daily living (IADL Lawton). From 8 issues, it allows to study the ability of the person to perform common activities: Ability to use the phone to go shopping, preparing food, do its housekeeping, to its activities bleaching, to use the means of transport, to ensure accountability in respect of salary and handle money.

SECONDARY OUTCOMES:
Consistency of the answers to each question of the IADL questionnaires between the two methods of administration | 1 month
  To assess the reliability of the collection of the questionnaire by phone (agreement answers to each question on the IADL), the secondary endpoint will be considered:
  - The consistency of the answers to each question of the IADL questionnaires between the two methods of administration: during the face-to-face interview, and by phone.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hôpital Charpennes - Memory Research Centre Lyon, Clinical Research Centre (CVF), Villeurbanne, France

REFERENCES:
- [Result] Dauphinot V, Boublay N, Moutet C, Achi S, Bathsavanis A, Krolak-Salmon P. Comparison of Instrumental Activities of Daily Living assessment by face-to-face or telephone interviews: a randomized, crossover study. Alzheimers Res Ther. 2020 Mar 13;12(1):24. doi: 10.1186/s13195-020-00590-w. PMID 32169093